CLINICAL TRIAL: NCT04924543
Title: OPtical Diagnosis Training to Improve Dysplasia Characterisation in Inflammatory Bowel Disease
Brief Title: OPtical Diagnosis Training to Improve Dysplasia Characterisation in IBD
Acronym: OPTIC-IBD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Birmingham (Other)
Collaborators: University of Calgary (Other); University of Milan (Other); Federico II University (Other); University of Bari Aldo Moro (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: ERN-18-0222A; REB21-0409 (Other: University of Calgary, Canada)
Record Dates: First submitted 2021-06-07; First posted 2021-06-14 (Actual); Last update posted 2022-05-18 (Actual); Status verified 2022-05

CONDITIONS: Inflammatory Bowel Diseases; Dysplasia Colon; Dysplasia, Crohn Disease-Associated; Polyp of Colon; Ulcerative Colitis; Crohn Colitis; Crohn Disease
Keywords: Endoscopy; Optical diagnosis; Dysplasia surveillance; Inflammatory bowel disease
MeSH Terms: conditions — Inflammatory Bowel Diseases; Colonic Polyps; Colitis, Ulcerative; Crohn Disease

STUDY DESIGN:
Intervention Model Description: All enrolled participants are allocated to the same intervention, with pre-course and post-course assessments.
  Participants will then be randomized 1:1 to one of two arms: (1) to receive short refresher training on optical diagnosis, or (2) no additional intervention.
  All participants will complete a final late post-course assessment to test knowledge retention from the training module and the impact of refresher training.
Masking Description: No masking planned
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Received short refresher training on optical diagnosis (Active Comparator): All participants receive access to the training module, with assessments at baseline, week 2 and week 8-12 Half of participants randomized 1:1 will also receive access to brief refresher training by week 8
  Interventions: Other: Online self-learning training module; Other: Refresher training
- No refresher training (Active Comparator): All participants receive access to the training module, with assessments at baseline, week 2 and week 8-12 This arm does not also receive access to brief refresher training
  Interventions: Other: Online self-learning training module

INTERVENTIONS:
Other: Online self-learning training module — Training module in optical diagnosis of IBD-associated dysplastic lesions during gastrointestinal endoscopy
Other: Refresher training — Brief refresher training in optical diagnosis of IBD-associated dysplastic lesions during gastrointestinal endoscopy
  Arms: Received short refresher training on optical diagnosis

SUMMARY:
People with inflammatory bowel diseases (IBD) can be at higher risk of developing abnormal areas in their bowel. These abnormal areas can be due to active inflammation, healed inflammation, polyps or pre-cancerous changes ("dysplasia"). It is for this reason that people with IBD are offered periodic surveillance colonoscopy procedures to identify, characterize and where necessary remove abnormal areas or lesions from the bowel. These can be difficult to characterize correctly, which is important to make the correct endoscopic diagnosis and management plan. Technical advancements in endoscopy mean that more tools are available to identify and characterize these lesions in real time during colonoscopy. Specialists regularly performing gastrointestinal endoscopy and colonoscopy ("endoscopists") will often receive special training, both during their initial postgraduate training and through continuous professional development programs.

This study aims to evaluate whether an online training platform can improve the ability of endoscopists to characterize dysplasia in IBD. The goal is to support improved decision-making during IBD surveillance, reporting of dysplastic lesions, and ultimately the care and outcomes of people with IBD.

DETAILED DESCRIPTION:
This study aims to evaluate whether an online training platform can improve the ability of endoscopists to characterise dysplasia in inflammatory bowel disease (IBD), to ultimately improve decision-making, reporting of dysplastic lesions and management during IBD surveillance.

Colonoscopy (endoscopic examination of the lower bowel) is a well-established screening tool to identify lesions within the bowel and objectively assess the degree of inflammation present. Patients with IBD, both Ulcerative colitis (UC) and Crohn's disease (CD), have a higher risk of developing cancers of the bowel and it is for this reason that they undergo regular surveillance procedures. Guidelines recommend surveillance procedures using high definition white light endoscopy alongside either Dye-Based Chromoendoscopy (DCE) or Virtual Chromoendoscopy (VCE), with targeted biopsies. However, the real world adoption of DCE and VCE is still modest. Due to technological advances there are alternative endoscopic imaging techniques that selectively enhance certain mucosal and vascular features, including narrow-band imaging (NBI), i-Scan optical enhancement (i-Scan-OE) and blue laser imaging (BLI).

These technologies have been demonstrated to be more effective than standard white light endoscopy. Despite these advances in technology, detecting dysplasia within areas of inflammation due to IBD is challenging. An endoscopic classification was recently developed by Iacucci M et al called "FACILE" to characterise in detail the mucosal and vascular pattern to predict histological colonic lesions in IBD. Since traditional lesion assessment systems such as (unmodified) Kudo pit pattern are less reliable in IBD, there is a need for a robust scoring system to assist clinicians in detecting and characterising lesions in IBD.

This project is to validate a training module on surveillance and colonic lesion characterisation in IBD. We aim to compare polyp detection in IBD surveillance procedures before and after training and evaluate the impact. As a sub-study, an additional randomisation process will take place whereby one group will receive additional focused top-up training and the other group will not. We will seek to compare the impact of feedback on knowledge retention.

Study stages:

* Stage 1. Potential participants are provided an electronic PIS outlining the study.
* Stage 2. Participants consent to the study and complete the pre-training assessment on REDCap (1 hour).
* Stage 3. Participants are provided with login details for online training.
* Stage 4. Participants complete the online training in their own time (1 hour).
* Stage 5. Participants complete the same assessment (as pre-training) and are given 1-2 weeks to complete this after training.
* Sub-study: Participants are randomised 1:1 to either receive or not receive a short refresher training module (15 min).
* Stage 6. After 8-12 weeks post-training participants are invited to complete the same assessment process (as pre-training).

All participants will receive computer-based training. Training will take place via an online computer- based self-learning platform. The training will include reviewing short videos of colorectal polyps in patients with IBD and videos of inflammation in IBD (quiescent, mild, moderate and severe) using NBI, i-Scan-OE and BLI. Patients were consented for the use of the use of videos for educational purposes. Videos used have been fully anonymised.

All Participants are given access to the secure REDCap platform hosted at the University of Birmingham. Participants will be required to register using a general survey to include their email address, anonymised demographic data, procedural experience and familiarity with optical endoscopic diagnosis platforms.

Participants comprise three categories: novice, training endoscopist and experienced endoscopist. The latter two are the key categories for evaluation.

* Novice will include medical students and junior doctors/residents who have previously had no or little endoscopic experience.
* Training endoscopists will be gastroenterology and general surgery trainees/residents/fellows.
* Experienced endoscopists will be fully qualified endoscopists such as GI and general surgery staff, consultants and nurse endoscopists.

Participants will then complete pre-training assessment prior to e-learning training. There are 26 video clips representative of different types of colonic lesions in IBD. Each video clip is typically 20-30 seconds. The overall duration of the assessment is around one hour.

Participants will then be given a login for the online training material and will complete this in their own time. Participants will be taught on endoscopic surveillance in IBD and how to characterise polyps accurately. The duration of the training module is 1 hour. It is interactive with optional components for tailored self-directed learning.

A post-training assessment will be completed in the next 1-2 weeks, using the same video clips, allowing us to compare the performance of participants before and after training. The assessment will be repeated after 8-12 weeks to assess the retention of skills.

An additional randomisation process on a 1:1 basis will take place, whereby one group will receive additional short refresher training following their responses to assessment questions and the other group will not. We will seek to compare the impact of feedback on sustainability of knowledge retention.

ELIGIBILITY:
Inclusion criteria:

* Specialist physicians performing gastrointestinal endoscopy
* Non-medical endoscopists
* Endoscopists in training with various levels of experience (such as Specialty Registrar, Fellow, Resident, non-medical endoscopists in training)
* Novice endoscopists with no or limited experience (no previous exposure bias to endoscopy training or practice)

Exclusion criteria:

* Unable to give informed consent to participate in study
* Unwilling to give informed consent to participate in study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 182 (Actual)
Dates: Start 2021-07-07 (Actual); Primary Completion 2021-12-20 (Actual); Study Completion 2022-04-30 (Actual)

PRIMARY OUTCOMES:
Change in percentage of participants who accurately characterized endoscopic lesions of the intestine in patients with inflammatory bowel disease - impact of training module | Baseline and 2 weeks
  Accuracy in characterization by modified SCENIC classification [Surveillance for Colorectal Endoscopic Neoplasia Detection and Management in Inflammatory Bowel Disease Patients: International Consensus Recommendations], modified Kudo pit pattern classification, FACILE classification [Frankfurt Advanced Chromoendoscopic Inflammatory Bowel Disease Lesions], optical prediction of final histopathological diagnosis

SECONDARY OUTCOMES:
Change in percentage of participants who accurately characterized endoscopic lesions of the intestine in patients with inflammatory bowel disease - impact of training module, impact of short refresher training | Baseline and 8-12 weeks
  Accuracy in characterization by modified SCENIC classification [Surveillance for Colorectal Endoscopic Neoplasia Detection and Management in Inflammatory Bowel Disease Patients: International Consensus Recommendations], modified Kudo pit pattern classification, FACILE classification [Frankfurt Advanced Chromoendoscopic Inflammatory Bowel Disease Lesions], overall optical prediction of final histopathological diagnosis
Change in percentage of participants who accurately characterized endoscopic lesions of the intestine in patients with inflammatory bowel disease - retention between participants randomized to receive or not receive refresher training | 2 weeks and 8-12 weeks
  Accuracy in characterization by modified SCENIC classification [Surveillance for Colorectal Endoscopic Neoplasia Detection and Management in Inflammatory Bowel Disease Patients: International Consensus Recommendations], modified Kudo pit pattern classification, FACILE classification [Frankfurt Advanced Chromoendoscopic Inflammatory Bowel Disease Lesions], overall optical prediction of final histopathological diagnosis
Change in participant assessment of confidence of prediction for each video (High vs. Low) - impact of training module | Baseline and 2 weeks
  Confidence in overall optical prediction of final histopathological diagnosis
Change in participant assessment of confidence of prediction for each video (High vs. Low) - impact of training module, impact of short refresher training | Baseline and 8-12 weeks
  Confidence in overall optical prediction of final histopathological diagnosis
Change in participant assessment of confidence of prediction for each video (High vs. Low) - at re-assessment between participants randomized to receive or not receive short refresher training | 2 weeks and 8-12 weeks
  Confidence in overall optical prediction of final histopathological diagnosis
Participant assessment of overall confidence in characterization of endoscopic lesions in patients with inflammatory bowel disease - impact of training module | Baseline assessment
  Confidence by Likert scale (0 = no confidence, 1, 2 , 3 = moderate confidence, 4, 5, 6 = high confidence)
Participant assessment of impact of training module on overall confidence in characterization of endoscopic lesions in patients with inflammatory bowel disease - impact of training module | Early post-training assessment at 2 weeks
  Confidence by Likert scale (0 = no confidence, 1, 2 , 3 = moderate confidence, 4, 5, 6 = high confidence)
Participant assessment of impact of training program on overall confidence in characterization of endoscopic lesions in patients with inflammatory bowel disease - impact of training module with or without brief refresher training | Late post-training assessment by 8-12 weeks
  Confidence by Likert scale (0 = no confidence, 1, 2 , 3 = moderate confidence, 4, 5, 6 = high confidence)

OTHER OUTCOMES:
Quality of training module | Baseline assessment
  Participant assessment of quality of each video (High vs. Low)
Quality of training module | Early post-training assessment by 2 weeks
  Participant assessment of quality of each video (High vs. Low)
Quality of training module | Late post-training assessment by 8-12 weeks
  Participant assessment of quality of each video (High vs. Low)
Quality of training module | At provision of training module by 2 weeks
  Module evaluation by Likert scales (strongly agree, agree, neither agree or disagree, disagree, strongly disagree) for "The module has been effective in helping me to learn" and "The module content was relevant" and "The module length was appropriate" and "I would recommend the module" and "The assessments matched the module content", and evaluation by free text comments "What have you learned in this module that will impact on your clinical practice?" and "Describe the best and worst thing about this module" and "How would you change or improve this module?"
Quality of brief refresher training | At provision of brief refresher training by 8 weeks
  Module evaluation by Likert scales (strongly agree, agree, neither agree or disagree, disagree, strongly disagree) for "The refresher training has been effective in helping me to consolidate my learning" and "The refresher training content was relevant" and "The refresher training length was appropriate" and "I would recommend including refresher training in the program", and evaluation by free text comments "Describe the best and worst thing about this refresher training" and "How would you change or improve this refresher training?"

CONTACTS AND LOCATIONS:
Overall Officials: Marietta Iacucci, MD PhD, Study Director — University of Birmingham; Jose G Ferraz, MD PhD, Principal Investigator — University of Calgary; Gian E Tontini, MD PhD, Principal Investigator — University of Milan
Locations (5):
- University of Calgary, Calgary, Alberta, Canada
- Italy (3):
  - University Aldo Moro, Bari
  - University of Milan, Milan
  - University Federico II, Napoli
- University of Birmingham, Birmingham, United Kingdom

IPD SHARING:
Plan to Share IPD: No
No plan to share IPD as not applicable to this study

REFERENCES:
- [Background] Clarke WT, Feuerstein JD. Colorectal cancer surveillance in inflammatory bowel disease: Practice guidelines and recent developments. World J Gastroenterol. 2019 Aug 14;25(30):4148-4157. doi: 10.3748/wjg.v25.i30.4148. PMID 31435169
- [Background] Bye WA, Ma C, Nguyen TM, Parker CE, Jairath V, East JE. Strategies for Detecting Colorectal Cancer in Patients with Inflammatory Bowel Disease: A Cochrane Systematic Review and Meta-Analysis. Am J Gastroenterol. 2018 Dec;113(12):1801-1809. doi: 10.1038/s41395-018-0354-7. Epub 2018 Oct 23. PMID 30353058
- [Background] Gabbani T, Manetti N, Bonanomi AG, Annese AL, Annese V. New endoscopic imaging techniques in surveillance of inflammatory bowel disease. World J Gastrointest Endosc. 2015 Mar 16;7(3):230-6. doi: 10.4253/wjge.v7.i3.230. PMID 25789093
- [Background] Iacucci M, McQuaid K, Gui XS, Iwao Y, Lethebe BC, Lowerison M, Matsumoto T, Shivaji UN, Smith SCL, Subramanian V, Uraoka T, Sanduleanu S, Ghosh S, Kiesslich R. A multimodal (FACILE) classification for optical diagnosis of inflammatory bowel disease associated neoplasia. Endoscopy. 2019 Feb;51(2):133-141. doi: 10.1055/a-0757-7759. Epub 2018 Dec 12. PMID 30541154
- [Background] Cassinotti A, Fociani P, Duca P, Nebuloni M, Davies SEC, Sampietro G, Buffoli F, Corona A, Maconi G, Ardizzone S. Modified Kudo classification can improve accuracy of virtual chromoendoscopy with FICE in endoscopic surveillance of ulcerative colitis. Endosc Int Open. 2020 Oct;8(10):E1414-E1422. doi: 10.1055/a-1165-0169. Epub 2020 Sep 22. PMID 33015345
- [Background] Mazzuoli S, Guglielmi FW, Antonelli E, Salemme M, Bassotti G, Villanacci V. Definition and evaluation of mucosal healing in clinical practice. Dig Liver Dis. 2013 Dec;45(12):969-77. doi: 10.1016/j.dld.2013.06.010. Epub 2013 Aug 7. PMID 23932331
- [Background] Vuitton L, Peyrin-Biroulet L, Colombel JF, Pariente B, Pineton de Chambrun G, Walsh AJ, Panes J, Travis SP, Mary JY, Marteau P. Defining endoscopic response and remission in ulcerative colitis clinical trials: an international consensus. Aliment Pharmacol Ther. 2017 Mar;45(6):801-813. doi: 10.1111/apt.13948. Epub 2017 Jan 23. PMID 28112419
- [Background] van der Laan JJH, van der Waaij AM, Gabriels RY, Festen EAM, Dijkstra G, Nagengast WB. Endoscopic imaging in inflammatory bowel disease: current developments and emerging strategies. Expert Rev Gastroenterol Hepatol. 2021 Feb;15(2):115-126. doi: 10.1080/17474124.2021.1840352. Epub 2020 Oct 31. PMID 33094654
- [Background] Iacucci M, Daperno M, Lazarev M, Arsenascu R, Tontini GE, Akinola O, Gui XS, Villanacci V, Goetz M, Lowerison M, Lethebe BC, Vecchi M, Neumann H, Ghosh S, Bisschops R, Kiesslich R. Development and reliability of the new endoscopic virtual chromoendoscopy score: the PICaSSO (Paddington International Virtual ChromoendoScopy ScOre) in ulcerative colitis. Gastrointest Endosc. 2017 Dec;86(6):1118-1127.e5. doi: 10.1016/j.gie.2017.03.012. Epub 2017 Mar 18. PMID 28322774
- [Background] Ibraheim H, Dhillon AS, Koumoutsos I, Gulati S, Hayee B. Curriculum review: colorectal cancer surveillance and management of dysplasia in IBD. Frontline Gastroenterol. 2018 Oct;9(4):271-277. doi: 10.1136/flgastro-2017-100919. Epub 2018 Feb 10. PMID 30245789
- [Background] Allen JE, Vennalaganti P, Gupta N, Hornung B, Choudhary A, Titi M, Alsop BR, Lim D, Sharma P. Randomized Controlled Trial of Self-directed Versus In-Classroom Education of Narrow Band Imaging in Diagnosing Colorectal Polyps Using the NICE Criteria. J Clin Gastroenterol. 2018 May/Jun;52(5):413-417. doi: 10.1097/MCG.0000000000000791. PMID 28945617
- [Background] Khan T, Cinnor B, Gupta N, Hosford L, Bansal A, Olyaee MS, Wani S, Rastogi A. Didactic training vs. computer-based self-learning in the prediction of diminutive colon polyp histology by trainees: a randomized controlled study. Endoscopy. 2017 Dec;49(12):1243-1250. doi: 10.1055/s-0043-116015. Epub 2017 Aug 14. PMID 28806820
- [Background] Smith SCL, Saltzman J, Shivaji UN, Lethebe BC, Cannatelli R; Birmingham Colonic Polyp Characterisation Group; Ghosh S, Iacucci M. Randomized controlled study of the prediction of diminutive/small colorectal polyp histology using didactic versus computer-based self-learning module in gastroenterology trainees. Dig Endosc. 2019 Sep;31(5):535-543. doi: 10.1111/den.13389. Epub 2019 Apr 8. PMID 30844114
- [Derived] Iacucci M, Bonovas S, Bazarova A, Cannatelli R, Ingram RJM, Labarile N, Nardone OM, Parigi TL, Piovani D, Siau K, Smith SCL, Zammarchi I, Ferraz JGP, Fiorino G, Kiesslich R, Panaccione R, Parra-Blanco A, Principi M, Tontini GE, Uraoka T, Ghosh S; OPTIC-IBD Study Group. Validation of a new optical diagnosis training module to improve dysplasia characterization in inflammatory bowel disease: a multicenter international study. Gastrointest Endosc. 2024 May;99(5):756-766.e4. doi: 10.1016/j.gie.2023.11.018. Epub 2023 Nov 21. PMID 37993058